CLINICAL TRIAL: NCT02806596
Title: Use of Bispectral Index to Guide Intubation During Sevoflurane Anesthesia in Children
Brief Title: Bispectral Index to Guide Intubation in Pediatric Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Claude Hallet, Chief of Clinic, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BIS02ch
Record Dates: First submitted 2016-06-08; First posted 2016-06-20 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sevoflurane (Other): * induction of anesthesia using sevoflurane administered with facial mask at inspired concentration of 6% (in a mixture of oxygen and nitrous oxyde)
  * intervention : titration of inspired sevoflurane concentration until targeted bispectral index
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — After at least 4 minutes of stable inspired sevoflurane concentration, that concentration will be titrated to obtain a targeted bispectral index (BIS) level required for perform laryngoscopy. This level was initially set at 40, based on a preliminary study showing that such level of BIS was obtained at the laryngoscopy after common general anesthesia induction. For the next patients, BIS target was set according to a sequential allocation method (up and down).

SUMMARY:
This prospective study aimed to determine the minimal level of Bispectral index needed for quality laryngoscopy before ear, nose and throat surgery in children.

DETAILED DESCRIPTION:
* Children will received intra-rectal premedication based on midazolam 0.4mg
* Children will be monitored according to standard guidelines
* One blinded anesthesiologist will be in charge of anesthesia induction and the other one will be in charge of data collection (end tidal sevoflurane concentration, sevoflurane minimal alveolar concentration, bispectral index) and guidance of induction according to the predetermined bispectral index (up and down allocation)

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiology physical status classification system :1 or 2
* scheduled ear, nose and throat surgery in a one day program
* oral intubation required

Exclusion Criteria:

* parents refusal
* recent respiratory infection
* epilepsy
* suspected difficult intubation

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
laryngeal conditions of intubation | 5 minutes
  specific conditions will be assessed and scored : jaw relaxation, vocal cord position, cough at intubation

IPD SHARING:
Plan to Share IPD: No
data will not been shared